CLINICAL TRIAL: NCT02162862
Title: Treating Disrupted Sleep in Individuals With Inflammatory Bowel Disease: A Novel Adjunctive Therapy for Chronic Inflammatory Illness
Brief Title: Treating Disrupted Sleep in Individuals With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eva Szigethy (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor-Investigator, Eva Szigethy, Associate Professor of Psychiatry, Pediatrics, and Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CCFA 13050045
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-06

CONDITIONS: Sleep Disturbance; Fatigue; Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Physical Illness; Wellbutrin
MeSH Terms: conditions — Parasomnias; Fatigue; Inflammatory Bowel Diseases | interventions — Behavior Therapy; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral Counseling (Other): Brief Behavioral Therapy for Sleep Disruption in IBD (BBTS-I). This treatment phase focuses on treating insomnia, a nighttime component of sleep disturbance delivered in 1:1 sessions which can be completed in person or by phone, except for initial session.
  Interventions: Behavioral: Behavioral Counseling
- Behavioral counseling + bupropion-SR (Other): Brief Behavioral Therapy for Sleep Disruption in IBD (BBTS-I) plus bupropion-SR (bupropion-Sustained Release). 8-week trial of bupropion-SR (target dose: 200-300 mg/day). bup-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement-sleep (REM) in medically ill populations.
  Interventions: Behavioral: Behavioral Counseling; Drug: bupropion-SR
- Healthy Control (No Intervention): The healthy control group includes individuals who are free of physical and psychiatric illness between the ages of 15-30.

INTERVENTIONS:
Behavioral: Behavioral Counseling
  Arms: Behavioral Counseling; Behavioral counseling + bupropion-SR
Drug: bupropion-SR
  Other Names: Wellbutrin
  Arms: Behavioral counseling + bupropion-SR

SUMMARY:
The purpose of this study is to determine if either a targeted type of talk therapy (Phase I) or medication, Wellbutrin, (Phase II) improve sleep disturbance and/or fatigue in individuals with Inflammatory Bowel Disease (IBD).

DETAILED DESCRIPTION:
The present study, sponsored by the Crohn's and Colitis Foundation of America, intends to provide information about the feasibility and effectiveness of treatments designed to lessen fatigue and improve sleep among youth with Crohn's disease (CD). Obtaining good sleep is vital in leading a healthy life. For youth with Inflammatory Bowel Disease (IBD), good sleep is key as patients are psychically and psychologically developing and maturing. Previous work suggests that 42% of youth with CD experience poor sleep: difficulty falling asleep, disruption in sleep, early morning awakening, or an absence of feeling refreshed after sleep. Poor sleep can negatively affect ones physical health, mental health, and stress level - each minimizing ones quality of life.

Participants in the study range from 15-30 years old, live with CD, and experience sleep disturbances, targeting 100 participants. Additionally, a healthy control group, 30 participants, is included for comparison. The study contains two phases and takes place over a 12-week period. Phase one involves partaking in 3-8 sessions of Brief Behavioral Therapy for Sleep in IBD (BBTS-I) with study clinician. The treatment teaches self-management techniques and sleep interventions through self-hypnosis/relaxation and reflection. After the treatment, participants are reevaluated. Those who respond well to the treatment are offered 1-2 booster sessions, those who do not show improvement move on to phase two.

In phase two, participants are offered an 8-week course of bupropion-sustained release (BUP-SR). BUP-SR reduces fatigue, depression, and inflammation, and enhances REM sleep. The prescribed dosage will increase from 100mg to 300 mg (150 mg 2x a day). Participant's characterization measures are assessed at the start, midpoint, and finish of the study to measure changes in sleep, fatigue, and mood. Also at these times, blood work is done in hopes of gaining an understanding of the cause of CD. At each of the three assessments, participants are asked to wear a wristwatch device for 7 days that records: total sleep time, wakefulness, and daytime information on napping and sleep hygiene. In addition, participants are asked to keep a brief sleep diary for a 7-day period. This study hopes to provide new treatments to increase the quality of life, primarily by improving sleep in patients with CD.

ELIGIBILITY:
Inclusion Criteria:

* IBD Group:

  * Biopsy confirmed Crohn's Disease
  * Qualifying scores on Multidimensional Fatigue Inventory and Pittsburgh Sleep Quality Index
* Healthy Volunteer Group:

  * Does not meet any exclusion criteria

Exclusion Criteria:

* IBD Group:

  * Meeting criteria for active alcohol or substance abuse or dependence
  * Current ongoing treatment with Wellbutrin
  * Females who are pregnant or plan to become pregnant within three months
  * Sleep disorder such as apnea, restless leg syndrome or use of Continuous positive airway pressure therapy (C-PAP)/Bilevel positive airway pressure (Bi-PAP)
  * Current IBD flare requiring hospitalization with intravenous steroid treatment
  * Other acute medical conditions or a history of chronic inflammatory condition other than IBD
  * Hemoglobin <10 with age and gender adjustments
  * History of seizure disorder
  * Acute infection within seven days
* Healthy Volunteer Group:

  * History or current episode of psychiatric disorder by Diagnositic and Statistical Manual (DSM-IV)
  * Current ongoing treatment with psychoactive medications
  * Medications for sleep in previous two weeks
  * Females who are pregnant or plan to become pregnant within three months
  * History of IBD, epilepsy, rheumatoid arthritis, lupus
  * Sleep disorder such as apnea, restless leg syndrome or use of Continuous positive airway pressure therapy (C-PAP)/Bilevel positive airway pressure (Bi-PAP)

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Presbyterian University Hospital of UPMC, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the Digestive Disorders Clinic at Presbyterian Hospital in Pittsburgh, PA. Recruitment began 11/13/13 and ended 2/18/16.
Groups:
- Healthy Control: The healthy control group included individuals who were free of physical and psychiatric illness between the ages of 15-30.
- Behavioral Counseling: Brief Behavioral Therapy for Sleep Disruption in IBD (BBTS-I). This treatment phase focuses on treating insomnia, a nighttime component of sleep disturbance delivered in 1:1 sessions which can be completed in person or by phone, except for initial session.
  Behavioral Counseling
  Within this arm, some participants offered bupropion-SR (bupropion-Sustained Release). 8-week trial of bupropion-SR (target dose: 200-300 mg/day). bup-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement-sleep (REM) in medically ill populations.
  bupropion-SR
- Behavioral Counseling + Bupropion: Brief Behavioral Therapy for Sleep Disruption in IBD (BBTS-I) plus bupropion-SR (bupropion-Sustained Release). 8 -week trial of bupropion-SR (target dose: 200-300mg/day). Bupropion-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement sleep (REM) in medically ill populations.
Period: Overall Study
Arm/Group | Healthy Control | Behavioral Counseling | Behavioral Counseling + Bupropion
Started | 31 | 35 | 33
Completed | 31 | 24 | 29
Not Completed | 0 | 11 | 4
Not completed — Lost to Follow-up | 0 | 11 | 0
Not completed — Subject did not feel the med was needed | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Counseling: Brief Behavioral Therapy for Sleep Disruption in IBD (BBTS-I). This treatment phase focuses on treating insomnia, a nighttime component of sleep disturbance delivered in 1:1 sessions which can be completed in person or by phone, except for initial session.
  Behavioral Counseling
- Control Group: Individuals free of physical and psychiatric illness.
- Behavioral Counseling + Bupropion: Brief Behavioral Therapy for Sleep Disruption in IBD (BBTS-I) plus bupropion-SR (bupropion-Sustained Release). 8-week trial of bupropion-SR (target dose: 200-300 mg/day). bup-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement-sleep (REM) in medically ill populations.
- Total: Total of all reporting groups
Arm/Group | Behavioral Counseling | Control Group | Behavioral Counseling + Bupropion | Total
Number analyzed (Participants) | 35 | 31 | 33 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 6 | 5 | 15
  Between 18 and 65 years | 31 | 25 | 28 | 84
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (4.7) | 23.5 (4.3) | 23.96 (5.76) | 23.7 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 19 | 60
  Male | 13 | 12 | 14 | 39
Region of Enrollment [Number; unit: participants]
  United States | 35 | 31 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Multidimensional Fatigue Inventory (MFI) for Each Arm
Description: MFI score range is 0-100. Higher score indicates higher level of fatigue.
Time Frame: Baseline (week 0) to end of study (week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Behavioral Counseling + Bupropion: 8-week trial of bupropion-SR (target dose: 200-300 mg/day). bup-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement-sleep (REM) in medically ill populations.
  bupropion-SR
Arm/Group | Behavioral Counseling | Healthy Control | Behavioral Counseling + Bupropion
Number analyzed (Participants) | 35 | 31 | 33
units on a scale | 18.727 (13.843) | -1.828 (5.8) | 16.367 (13.962)
Statistical Analysis 1: Comparison: Behavioral Counseling; Test type: Other; p < 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: Behavioral Counseling + Bupropion; Test type: Other; p < 0.005, t-test, 2 sided
Statistical Analysis 3: Comparison: Healthy Control; Test type: Other; p = .102, t-test, 2 sided

2. Primary Outcome: Change in Baseline in Pittsburgh Sleep Quality Index (PSQI) for Each Arm
Description: PSQI score range is 0-21 with higher score indicating greater sleep disturbance.
Time Frame: Baseline (week 0) to end of study (week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Behavioral Counseling + Bupropion: Within this arm, some participants offered bupropion-SR (bupropion-Sustained Release). 8-week trial of bupropion-SR (target dose: 200-300 mg/day). bup-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement-sleep (REM) in medically ill populations.
  bupropion-SR
Arm/Group | Behavioral Counseling | Healthy Control | Behavioral Counseling + Bupropion
Number analyzed (Participants) | 35 | 31 | 33
units on a scale | 4.857 (3.928) | -.154 (1.69) | 6.571 (3.696)
Statistical Analysis 1: Comparison: Behavioral Counseling; Test type: Other; p < 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Control; Test type: Other; p = .646, t-test, 2 sided
Statistical Analysis 3: Comparison: Behavioral Counseling + Bupropion; Test type: Other; p < 0.005, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The study was conducted over a period of 2 years. Each subject participated in the study for 4 months. No adverse events were reported for any subjects during their time in the study.
Groups:
- Behavioral Counseling + Bupropion: Participants offered bupropion-SR (bupropion-Sustained Release). 8-week trial of bupropion-SR (target dose: 200-300 mg/day). Bup-SR, a noradrenergic dopaminergic reuptake inhibitor (NDRI). NDRI has been shown to improve fatigue and rapid eye movement-sleep (REM) in medically ill populations.
Arm/Group | Healthy Control | Behavioral Counseling | Behavioral Counseling + Bupropion
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/35 | 0/33

LIMITATIONS AND CAVEATS:
There were no limitations to this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No